CLINICAL TRIAL: NCT06509815
Title: Safety, Feasibility, and Efficacy of a Bio-experiential Intervention, Multi-sensory Intervention Room Application (MIRA), During Neurosciences ICU Stay
Brief Title: Multi-sensory Intervention Room Application (MIRA) Device in the NSICU
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Neha Dangayach, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY-23-00967
Record Dates: First submitted 2024-05-02; First posted 2024-07-19 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Post Intensive Care Syndrome
Keywords: Post Intensive Care Syndrome; Bio-Experiential Space; Biophilic Design
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MIRA in the NSICU (Experimental): The Intervention arm will experience the device, MIRA, during their stay in the NSICU.
  Interventions: Device: MIRA
- Control (No Intervention): The Control arm will not experience the device.

INTERVENTIONS:
Device: MIRA — The study device is a Multi-Sensory Stimulation Device named MIRA, which uses commercially available hardware and builds off the SOLUNA software created by Studio Elsewhere. The device produces audio and visual stimuli of immersive experiences. Participants in the intervention group will either have periodic or scheduled intervention sessions. The study team member will roll the MIRA device into the patient participant's room before the session and roll it out after. The intervention requires the participant to be in bed. The study team member will set up the device and start the intervention session which can last between 15-60 minutes. During the session, data will be collected by the study team member.
  Arms: MIRA in the NSICU

SUMMARY:
The purpose of this research study is to determine the safety, feasibility, and efficacy of a device, MIRA, on the physical, mental, and cognitive health of Neurosciences Intensive Care Unit (NSICU) patients.

The study device is a Multi-Sensory Stimulation Device named MIRA, which uses commercially available hardware and builds off the SOLUNA software created by Studio Elsewhere, which produces audio and visual immersive experiences. The current device, Model M1, is a prototype developed for sole investigational purposes of this study and is not commercially available.

Participants, who will be patients and staff of the NSICU, will complete questionnaires regarding safety, feasibility, and efficacy. The research team will enroll 20 patient and 15 staff participants. The trial is expected to last 12 months.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, an individual must meet all of the following criteria:

For NSICU Staff:

* Current employee at NSICU
* Aged >/= 18

For NSICU Patients:

* Currently admitted to the Mount Sinai Hospital NSICU for any diagnosis OR a Legally Authorized Representative (LAR) for the patient, and expected to stay for at least 48 hours
* Provision of signed and dated informed consent form (ICF)
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Aged >/= 18
* Any sex or gender identity
* Currently admitted to the Mount Sinai Hospital NSICU for any diagnosis OR a Legally Authorized Representative (LAR) for the patient, and expected to stay for at least 48 hours

Exclusion Criteria

* Not a Mount Sinai NSICU patient
* No LAR present and unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-08-25 (Actual); Primary Completion 2025-07-12 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM) | Within 2 days of the device used in the patient room during stay in ICU
  Implementation success will be assessed using the Acceptability of Intervention Measure (AIM). AIM is a 4-item measure used to determine the extent to which stakeholders (e.g., parents, providers, administrators) believe an intervention or implementation strategy is acceptable. Total score ranges from a minimum score 4 (unacceptable) to a maximum score 20 (very acceptable), with higher scores indicating greater acceptability of the intervention.
Intervention Appropriateness Measure (IAM) | Within 2 days of the device used in the patient room during stay in ICU
  Implementation success will be assessed using the Intervention Appropriateness Measure (IAM). IAM is a 4-item measure used to determine the extent to which stakeholders (e.g. parents, providers, administrators) believe an intervention or implementation strategy is appropriate or suitable for the situation. Total score ranges minimum 4 (unacceptable) to maximum 20 (very acceptable), with higher scores indicating greater appropriateness of the intervention strategy being evaluated.
Feasibility of Intervention Measure (FIM) | Within 2 days of the device used in the patient room during stay in ICU
  Implementation success will be assessed using the Feasibility of Intervention Measure (FIM). FIM is a 4-item measure used to determine the extent to which an intervention or implementation strategy is feasible to implement. Total score ranges from a minimum of 4 (not feasible) to a maximum of 20 (very feasible), with higher scores indicating greater perceived feasibility of the intervention strategy being evaluated.

SECONDARY OUTCOMES:
Intubated pain measured using Critical Care Pain Observation Tool | daily, average 4 days in ICU
  The Critical Care Pain Observation Tool (CCPOT) is an 8-item measure used to assess self-reported pain levels in intubated, critically ill patients who cannot self-report. Total CCPOT score ranges from a minimum of 0 (no pain behaviors observed) to a maximum of 8 (significant behaviors indicating severe pain), with higher scores indicating higher pain levels in intubated patients.
Non-intubated pain measured using Pain Scale | daily, average 4 days in ICU
  The Pain Scale is used to assess self-reported pain levels in critically ill patients who are not intubated and can self-report pain. Total score on the Pain Scale ranges from a minimum of 0 (no pain) to a maximum of 10 (worst/most severe pain), with higher scores indicating more intense pain levels in non-intubated patients.
Type of pain medication administration | daily, average 4 days in ICU
  Categorical information on the type of medication administered (sedatives, analgesics, anti-seizure medications, anti-hypertensives, pressors, antibiotics, antipsychotics, other)
Generalized Anxiety Disorder 7 Scale Score | Baseline, Day 0
  The Generalized Anxiety Disorder 7-item (GAD-7) scale is used to assess self-reported anxiety symptoms. Total GAD-7 score ranges from a minimum of 0 (no anxiety) to a maximum of 21 (severe anxiety), with higher scores indicating greater anxiety severity.
Generalized Anxiety Disorder 7 Scale Score | At Discharge, approximately 4 days
  The Generalized Anxiety Disorder 7-item (GAD-7) scale is used to assess self-reported anxiety symptoms. Total GAD-7 score ranges from a minimum of 0 (no anxiety) to a maximum of 21 (severe anxiety), with higher scores indicating greater anxiety severity.
Generalized Anxiety Disorder 7 Scale Score | Up to 6 months
  The Generalized Anxiety Disorder 7-item (GAD-7) scale is used to assess self-reported anxiety symptoms. Total GAD-7 score ranges from a minimum of 0 (no anxiety) to a maximum of 21 (severe anxiety), with higher scores indicating greater anxiety severity.
Patient Health Questionnaire 2 (PHQ2) Scale Score | Baseline, Day 0
  The Patient Health Questionnaire-2 (PHQ-2) is a 2-item screening tool used to assess depressed mood and anhedonia to screen for depression. PHQ-2 scores range from 0 to 6, with higher scores suggesting a higher likelihood of depression requiring further evaluation with the longer PHQ-9.
Patient Health Questionnaire 2 (PHQ2) Scale Score | At Discharge, approximately 4 days
  The Patient Health Questionnaire-2 (PHQ-2) is a 2-item screening tool used to assess depressed mood and anhedonia to screen for depression. PHQ-2 scores range from 0 to 6, with higher scores suggesting a higher likelihood of depression requiring further evaluation with the longer PHQ-9.
Patient Health Questionnaire 2 (PHQ2) Scale Score | Up to 6 months
  The Patient Health Questionnaire-2 (PHQ-2) is a 2-item screening tool used to assess depressed mood and anhedonia to screen for depression. PHQ-2 scores range from 0 to 6, with higher scores suggesting a higher likelihood of depression requiring further evaluation with the longer PHQ-9.
Patient Health Questionnaire 9 (PHQ9) Scale Score | Baseline, Day 0
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item self-report tool used to assess depression severity. PHQ-9 scores range from 0 to 27, with higher scores indicating more severe depressive symptoms.
Patient Health Questionnaire 9 (PHQ9) Scale Score | At Discharge, approximately 4 days
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item self-report tool used to assess depression severity. PHQ-9 scores range from 0 to 27, with higher scores indicating more severe depressive symptoms.
Patient Health Questionnaire 9 (PHQ9) Scale Score | Up to 6 months
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item self-report tool used to assess depression severity. PHQ-9 scores range from 0 to 27, with higher scores indicating more severe depressive symptoms.
Awareness of person, place, and time | Up to 6 months
  Neurological assessment used to assess mental status. Mental status checks if a person has awareness of person, place, and time.
Motor Status | Up to 6 months
  Neurological assessment used to asses motor status. Motor strength is ranked 0-5 (5 meaning full function) for both upper and lower extremities.
Response to noxious stimuli and/or touch | Up to 6 months
  Neurological assessment used to assess sensory status. Sensory status notes if the patient responds to noxious stimuli or not.
Insomnia Severity Index to measure sleep quality | Up to 6 months
  The Insomnia Severity Index (ISI) is a 7-item questionnaire used to assess perceived insomnia severity. ISI scores range from 0 to 28, with higher scores indicating more severe levels of insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Neha Dangayach, Principal Investigator — Principal Investigator
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No